CLINICAL TRIAL: NCT03402477
Title: "Watch and Wait" in Patients With Complete Clinical Response (cCR) After Neo-adjuvant Chemoradiotherapy for Primary Locally Advanced Rectal Cancer.
Brief Title: "Watch and Wait" After Neo-adjuvant Chemoradiotherapy for Primary Locally Advanced Rectal Cancer.
Acronym: NORWAIT
Status: Terminated | Type: Observational
Why Stopped: Suspicion of adverse events
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University Hospital of North Norway (Other); St. Olavs Hospital (Other); Helse-Bergen HF (Other); Sorlandet Hospital HF (Other Government); Oslo University Hospital (Other); University Hospital, Akershus (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUSID674
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer
Keywords: locally advanced, neo-adjuvant treatment, Watch & Wait
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among patients treated for locally advanced rectal cancer with neo-adjuvant radio-chemotherapy, about 15% will have complete clinical response in terms of no visible tumor or ulcerations on the site of the primary tumor, or whitening of the rectal wall or telangiectasia. In this Norwegian national multicenter observational study, patients with complete clinical response (cCR) after neo-adjuvant treatment for rectal cancer as defined by national guidelines, will be invited to a Watch&Wait program with a specially designed follow-up in order to see if the tumor has disappeared permanently, or if there is regrowth of the tumor. Primary endpoint is the true regrowth rate in an unselected national cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma of the rectum within 15 cm from the anal verge measured by rigid proctoscopy
* Patients who have completed neoadjuvant treatment according to national guidelines for rectal cancer, i.e., radiotherapy or chemo-radiotherapy (at least 40 Gy) or short-course radiotherapy combined with chemotherapy
* Patients aged ≥18 years of age are eligible for inclusion. However, patients aged ≤40 years are recommended to undergo surgery on the theoretical base of a possibly more aggressive tumour disease in this age group, and will be asked to participate in the study by consenting to recording of data. Those patients who insist on W&W approach after careful consideration and well-documented informed consent are eligible for entering the W&W protocol.
* Given informed consent
* Stage I-III rectal cancer; however, patients with limited liver metastases who undergo primary liver surgery as part of a "liver first" treatment approach may be included

Exclusion Criteria:

* Patients without cCR
* Patients unable to give informed consent
* Patients with short course radiotherapy (5x5 Gy) without additional chemotherapy, or patients receiving less than 40 Gy in long course CRT
* Patients with cCR but with increasing tumour growth on MRI after preoperative treatment
* Patients with metastatic disease at the time of diagnosis with the exception of those who are eligible for "liver first" treatment approach as part of an intention to cure approach.
* Patients previously diagnosed and treated for malignant disease in the pelvic region with radio- or chemoradiotherapy
* Other circumstances that may interfere with successful participation in the W&W protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in Norway with rectal cancer treated with neo-adjuvant radio-chemotherapy according to Norwegian national guidelines, who have complete clinical response at 6-12 weeks after fulfilled treatment
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Rate of regrowth | Baseline to 5 years
  rate of regrowth of tumor after initial complete clinical response (cCR) in patients who undergo a specially designed Watch & Wait program and without surgical removal of the rectum; to determine the positive predictive value of cCR.

SECONDARY OUTCOMES:
The rate of cCR after preoperative CRT | Baseline to 5 years
  To calculate the rate of cCR in an national unselected cohort
Metachronous distant metastases in patients following the W&W protocol | Baseline to 5 years
  To calculate the rate of the occurrence of distant metastases in patients who undergo the watch & Wait program
Overall and cancer-specific survival protocol compared to patients with ypCR, i.e. patients with complete pathologic response after resection. | Baseline to 5 years
  To analyse the overall and cancer-specific survival of patients with cCR following the W&W
Patient-reported outcome measures - rectal function (LARS) and quality of life (QoL) | Baseline to 5 years
  To evaluate the effect of the Watch and wait program on rectal function by using the Low anterior resection syndrome (LARS) score
Patient-reported outcome measures - quality of life (LARS) and quality of life (QoL) | Baseline to 5 years
  To measure the effect of the Watch and wait program on quality of life by using the EORTC QLQ C30
Sensitivity, specificity and overall diagnostic accuracy of MRI with regard to the diagnosis of complete response | Baseline to 5 years
  To compare the regression grade obtained by multi parametric MRI protocol to the clinical diagnose of complete response at baseline, i.e. clinical diagnosis of complete response
Diagnostic accuracy of MRI to detect regrowth during follow-up after complete response | Baseline to 5 years
  To compare the accuracy of multi parametric MRI protocol with clinical examination during follow-up with regard to possible regrowth of the tumour

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig Kørner, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (7):
- Norway (7):
  - Haukeland University Hospital, Bergen
  - Sørlandet Hospital Kristiansand, Kristiansand
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital Northern Norway, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No